CLINICAL TRIAL: NCT02164968
Title: Assessment of Respiratory Symptoms After Corticosteroid Treatment Period Using Impedance Pneumography
Acronym: IP-ASTMA_2
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University of Technology (Other)
Responsible Party: Principal Investigator, Jussi Karjalainen, MD, Tampere University Hospital
Other Study IDs: R14027
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Obstructive Bronchitis
Keywords: Device investigation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obstructive bronchitis: 1-5 year old patients who have visited the TAYS emergency room due to obstructive bronchitis and have been instructed to begin a three-month period of inhaled corticosteroid (ICS) treatment as per national guidelines.

SUMMARY:
INTRODUCTION

Lung function assessment of preschool children is hindered by their limited co-operation in conventional tests such as peak expiratory flow (PEF) or spirometry and the methods available for younger children are, again, laborious and time consuming. However, impedance pneumography (IP) records indices of airway obstruction during normal sleep at home and has been shown accurate in wheezy preschool children (Seppä et al. J Appl Physiol 2013).

AIM OF THE STUDY

The general purpose of this study is to assess the clinical value of the information provided by overnight home recording of tidal breathing by means of IP technique in young children with asthmatic symptoms and inhaled corticosteroid (ICS) medication.

The main hypothesis is that IP measurement can distinguish between groups whose asthmatic symptoms recur or do not recur after ending the ICS drug treatment period.

METHODS

The study recruits 1-5 year old children (n=75) who have presented at the emergency room due to obstructive bronchitis and for whom an ICS drug treatment period has been prescribed based on the national guidelines.

The subjects will perform three overnight IP measurements at home at two weeks intervals close to and after ending of the treatment period.

SIGNIFICANCE OF THE STUDY

Being an affordable, simple and convenient ambulatory measurement method, IP may bring needed objectivity to asthma diagnostics and asthma drug response assessment in young children.

DETAILED DESCRIPTION:
QUALITY CONTROL AND QUALITY ASSURANCE

Information of study personnel and training All personnel involved with the use of the IP measurement device will be instructed by Ville-Pekka Seppä.

Protocol amendments Essential amendments in the research protocol will be reviewed by the institutional review board and informed to National Supervisory Authority of Welfare and Health (Valvira).

DATA HANDLING AND RECORD KEEPING Electronic data collection Electronic data will consist of IP recorder device data files (.ipr). Upon complete protocol execution there will be three files for each patient. These files will be stored in a computer in TAYS Allergiakeskus.

Data management Access to all collected patient information and the patient information collected before the study in the primary care centers will be accessible to RN Tiina Mäki (0503439195), MD Marita Paassilta, and MD Jussi Karjalainen of Allergiakeskus.

Research group members from TUT will have access only to data that does not enable identifying individual patients and where individual patients are referred to by participant codes.

Study subject register The study subject register will be treated per the Finnish Personal Data Act article 10.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-5 yrs
* Recurrent obstructive bronchitis
* Inhaled corticosteroid treatment has been prescribed

Exclusion Criteria:

* Laryngeal disease
* Tracheobronchial malacia
* Parenchymal lung disease
* History of bronchopulmonary dysplasia
* Active implantable medical such as pacemakers

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 1-5 year old patients who have visited the TAYS emergency room due to obstructive bronchitis and have been instructed to begin a three-month period of inhaled corticosteroid (ICS) treatment as per national guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2014-05; Primary Completion 2017-11 (Actual); Study Completion 2020-03-27 (Actual)

PRIMARY OUTCOMES:
Ability of IP measurement to distinguish patient subgroups | 1 wk before to 4 weeks after end of ICS period
  Comparison of the measures derived from the IP measurement (the investigational device) between the subgroups in the cohort at three times: 1 wk before end of ICS period, 1-2 wk after ending ICS period, 3-4 wk after ending ICS period

CONTACTS AND LOCATIONS:
Overall Officials: Jussi Karjalainen, MD, Principal Investigator — Tampere University Hospital
Locations (2):
- Finland (2):
  - TAYS Allergiakeskus, Tampere
  - Tampere University of Technology / ELT Dept, Tampere

REFERENCES:
- [Background] Seppa VP, Pelkonen AS, Kotaniemi-Syrjanen A, Makela MJ, Viik J, Malmberg LP. Tidal breathing flow measurement in awake young children by using impedance pneumography. J Appl Physiol (1985). 2013 Dec;115(11):1725-31. doi: 10.1152/japplphysiol.00657.2013. Epub 2013 Oct 3. PMID 24092693